CLINICAL TRIAL: NCT03441490
Title: Internet-delivered Cognitive Behavioural Therapy for Adolescents With Anxiety: A Factorial Design
Brief Title: Internet-delivered Cognitive Behavioural Therapy for Adolescents With Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, professor Gerhard Andersson, Linkoeping University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2017/489-31.
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Anxiety
Keywords: Learning Support; Chat; Adolescents
MeSH Terms: conditions — Anxiety Disorders | interventions — Choline O-Acetyltransferase

STUDY DESIGN:
Intervention Model Description: Design is a two-by-two factorial randomized trial with four intervention groups: 1, ICBT with therapeutic guidance through mail. 2, ICBT with therapeutic guidance through chat. 3, ICBT with learning support and terapeutic guidance through mail. 4. ICBT with learning support and terapeutic guidance through chat.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICBT standard (Active Comparator): Internet-based cognitive behavioural therapy with therapeutic guidance through mail
  Interventions: Behavioral: Guided-ICBT for adolescents with anxiety
- ICBT chat (Experimental): Internet-based cognitive behavioural therapy with therapeutic guidance through chat
  Interventions: Behavioral: Guided-ICBT with chat
- ICBT learning support (Experimental): Internet-based cognitive behavioural therapy with learning support and therapeutic guidance through mail
  Interventions: Behavioral: Guided-ICBT with learning support
- ICBT with learning support and chat (Experimental): Internet-based cognitive behavioural therapy with learning support and therapeutic guidance through chat
  Interventions: Behavioral: Guided-ICBT with learning support and chat

INTERVENTIONS:
Behavioral: Guided-ICBT for adolescents with anxiety — Internet-based cognitive behavioural therapy with therapeutic guidance through mail, 8 weeks.
  Arms: ICBT standard
Behavioral: Guided-ICBT with chat — Internet-based cognitive behavioural therapy with therapeutic guidance through chat, 8 weeks.
  Arms: ICBT chat
Behavioral: Guided-ICBT with learning support — Internet-based cognitive behavioural therapy with learning support and therapeutic guidance through mail, 8 weeks.
  Arms: ICBT learning support
Behavioral: Guided-ICBT with learning support and chat — Internet-based cognitive behavioural therapy with learning support and therapeutic guidance through chat, 8 weeks.
  Arms: ICBT with learning support and chat

SUMMARY:
The purpose of this study is to evaluate the effects of learning support and chat on treatment outcome in internet-administrated cognitive behaviour therapy (ICBT) for adolescents with anxiety.

DETAILED DESCRIPTION:
The study is set up as a factorial design with two independent variables: 1: Learning support and 2: chat-sessions in real time. The intervention tested is based on cognitive behavior therapy delivered over the internet via a secure treatment platform. Participants in the study are recruited from the general public via social media. The intervention is in Swedish.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 15-19 years old
* Have symptoms of anxiety, anxiety disorder

Exclusion Criteria:

* Suicidal ideation
* Alcohol addiction
* other major primary psychiatric disorder
* Ongoing psychological treatment
* recent (during last 4 weeks) change in psychiatric medication

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures clinical anxiety. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Beck Depression Inventory - II (BDI-II) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures clinical depression. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire for Children (PSWQ - C) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures the tendency of youth to engage in excessive, generalized and uncontrollable worry. Respondents rates each item on a 4-point Likert scale consisting of never (0), sometimes (1), often (2) and always (3). The scores from each item are summed together to yield a total score that ranges from 0-42, with higher scores reflecting higher levels of worry. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Generalised Anxiety Disorder (GAD-7) | First week of treatment and then once a week during the treatment-period, two weeks post treatment, six months post treatment and 12 months post treatment.
  Measures severity of generalised anxiety.
Mini-Social Phobia Inventory (MINI-SPIN) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures clinical social phobia. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Agoraphobic Cognitions Questionnaire (ACQ) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures fearful cognitions associated with panic attacks and agoraphobia. The ACQ consists of 14 items which will be scored as a total scale in this study. worry. Respondents rates each item on a 5-point Likert scale consisting of never (1), Thought never occurs (2), Thought rarely occurs (3) Thought occurs during half of the times when I am nervous (4) Thought usually occurs (5) Thought always occurs when I am nervous. ACQ can be divided into two subscales: Loss of Control and Physical Concerns. Each of the subscales consists of 7 items.The total scores (or the subscales) are calculated by averaging the responses to the individual items composing that score. Higher scores indicates higher levels of fearful cognitions. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Satisfaction With Life Scale (SWLS) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures global cognitive judgements of one's life satisfacation as a whole, on a 5-item scale. Respondants rates how much they agree or disagree on a 7-pont scale ranging from (7) strongly agree to (1) strongly disagree, where higher scores indicates higher levels of life satisfaction. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Rosenberg Self-Esteem Scale (RSES) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Evaluates individual self-esteem. The scale is a ten item Likert scale with items answered on a four point scale, from (0) strongly agree to strongly disagree (3), where higher scores indicates higher self-esteem. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Alcohol Use Disorders Identification Test (AUDIT) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  Measures alcohol consumption, drinking behaviors, and alcohol-related problems. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Knowledge of CBT strategies (developed by the research group) | Two weeks pre treatment, two weeks post treatment, six months post treatment and 12 months post treatment
  A brief 16-item questionnaire that measures explicit, declarative knowledge about core CBT-principles and therapeutic points. Higher scores indicates more knowledge. Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden